CLINICAL TRIAL: NCT02414152
Title: A Phase I & II Open-label Study of the Effects of Anakinra (Kineret) in Corticosteroid-resistant Subjects With Sudden Sensorineural Heaing Loss (SSNHL)
Brief Title: Study of the Effects of Anakinra in Corticosteroid-resistant Subjects With Sudden Sensorineural Hearing Loss
Acronym: SSNHL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Early study termination occurred due to inability to secure funding
Sponsor: Andrea Vambutas (Other)
Responsible Party: Sponsor-Investigator, Andrea Vambutas, Chair, Department of Otolaryngology and Communicative Disorders, Northwell Health
Organization: Northwell Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-333B
Record Dates: First submitted 2015-02-23; First posted 2015-04-10 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Hearing Loss, Sudden
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anakinra (Experimental): 100mg of Anakinra administered as a daily subcutaneous injection
  Interventions: Drug: anakinra

INTERVENTIONS:
Drug: anakinra — 100mg of anakinra adminstered by a subcutaneous injection for a minimum of 28 days, retreatment with additional 28 day cycle based on clinical response
  Other Names: Kineret

SUMMARY:
The purpose of this study is to determine if anakinra (an interleukin-1 receptor antagonist) can improve hearing thresholds in patients with sudden sensorineural hearing loss that did not respond to oral steroid therapy. The patients to be enrolled will have recently completed a course of oral steroids and demonstrated no change in their audiometric thresholds following corticosteroid therapy.

The investigators will be measuring hearing thresholds (Pure tone average and word recognition scores) before and after anakinra and correlating these findings with circulating IL-1 levels in the patient's blood.

DETAILED DESCRIPTION:
For patients that experience an acute, sensorineural decline in hearing, timely corticosteroid administration may result in preservation of some or all of the hearing. For patients with sudden sensorineural hearing loss who have failed to respond to corticosteroid therapy, this study will be offered to determine if anakinra is a safe and effective alternative therapy for clinical hearing restoration. The investigators have previously demonstrated that IL-1beta inhibition (with anakinra) in a small cohort of patients with steroid resistant autoimmune inner ear disease was effective in demonstrating audiological improvements.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have Sudden Sensorineural Hearing Loss in one ear, with a no greater than 25 dB PTA in the contralateral ear.
2. Age and Gender: male and female subjects, age ≥ 18 but ≤ 75, will be recruited.
3. Patients must be capable of understanding and giving informed consent.
4. Patients must have SNHL of greater than or equal to 30dB at three contiguous frequencies in one ear which evolved in three days or less, with a PTA of 25dB or less in the contralateral ear.
5. Patients must have previously undergone a trial of high-dose corticosteroid therapy, at 60 mg daily for a minimum of seven days, with a variable taper thereafter that consists of a total of 14 consecutive days of corticosteroid use. Patients must have demonstrated less than a 5 decibel average improvement in their PTA in response to corticosteroids as measured by their audiogram.
6. NO greater than 30 days may elapse from the discontinuation from the initial course of steroid treatment to the time of enrollment.

Exclusion Criteria:

1. Patients over 75 years of age, because there is a higher incidence of infections in the elderly population in general, caution should be used in treating the elderly.
2. Patients with evidence of retrocochlear pathology (vestibular schwannoma) or inner ear malformation (Mondini Malformation or Enlarged Vestibular Aqueduct) based on imaging.
3. Patients concurrently receiving methotrexate or TNF-antagonist therapy.
4. Patients with a diagnosis of any immunodeficiency syndrome.
5. Patients with active or chronic infections.
6. Patients currently receiving, or having received treatment for a malignancy in the past three years.
7. Patients with a diagnosis of chronic renal insufficiency (a creatinine clearance of <49mL/min) or chronic renal failure.
8. Patients with evidence of neutropenia (an ANC of <1000) prior to treatment with anakinra.
9. Known hypersensitivity to E. coli derived products.
10. Latex sensitivity.
11. Any patient that received a live vaccine < 3 months prior to enrollment.
12. Any patient with a history of active narcotic abuse, including prescription narcotics.
13. Pregnant or lactating females.
14. Children, < age 18
15. .Non-English speaking patients, as the word recognition scoring is in English and is a vital component to the efficacy analysis.
16. Any patient that tests positive for Hepatitis B, C, HIV or tuberculosis on screening, with the exception of presence of antibodies to Hepatitis B in subjects reporting prior vaccination, and presence of positive skin testing for TB in subjects who received BCG in the past.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Vambutas, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore-LIJ Hearing and Speech Center, New Hyde Park, New York, United States

REFERENCES:
- [Result] Vambutas A, Lesser M, Mullooly V, Pathak S, Zahtz G, Rosen L, Goldofsky E. Early efficacy trial of anakinra in corticosteroid-resistant autoimmune inner ear disease. J Clin Invest. 2014 Sep;124(9):4115-22. doi: 10.1172/JCI76503. Epub 2014 Aug 18. PMID 25133431

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anakinra
Started | 2
Completed | 0 (Both subjects completed 56 days of anakinra but did not complete all visits in observational period)
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anakinra
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Response to Anakinra in Corticosteroid Resistant Patients With SSNHL
Description: Patients who had a response to anakinra based on hearing threshold improvement compared to their pre-treatment threshold.
Time Frame: 120 days
Population: Zero subjects were analyzed because both enrolled subjects were withdrawn after receiving 56 days of anakinra because no hearing improvement was noted. They did not complete the entire study.
Arm/Group | Anakinra
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Anakinra
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anakinra (N=2)
injection site reaction (Skin and subcutaneous tissue disorders) | 2
headache (Nervous system disorders) | 1
fatigue (General disorders) | 1
leg edema (Vascular disorders) | 1 — Slight lower leg pitting edema noted 1 months after study injections started- resolved after 1 week
dermatitis (Skin and subcutaneous tissue disorders) | 1 — Subject noted arms were very itchy after trip to Cayman Islands- resolved in 3 days
increased tinnitus (Ear and labyrinth disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination of the study secondary to inability to secure funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No